CLINICAL TRIAL: NCT05140304
Title: Quantitative and Qualitative Analysis of Foveal Avascular Zone Characteristics in Different Stages of Diabetic Retinopathy Using Optical Coherence Tomography Angiography (OCT-A)
Brief Title: Analysis of FAZ in Diabetic Retinopathy Using OCT Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kareem Mohammad Ali (Other)
Responsible Party: Sponsor-Investigator, Kareem Mohammad Ali, Resident, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OCT angiography
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A (Other)
  Interventions: Device: OCT angiography

INTERVENTIONS:
Device: OCT angiography — OCT angiography of foveal avascular zone in diabetic retinopathy

SUMMARY:
Study and assessment of characteristic changes in foveal avascular zone during different stages of diabetic retinopathy using OCTA.

DETAILED DESCRIPTION:
OCTA is superior to other retinal imaging techniques like fluorescein angiography(FA) as it does not require dye injection, Intravenous dye injection is time consuming and can have adverse side effects. Furthermore, the edges of the capillaries can become blurred due to dye leakage and imaging of the retina can only be 2D when using FA.

OCTA provides both structural and functional (i.e. blood flow) information in tandem. The "corresponding" OCT b-scans can be co-registered with the simultaneous OCT angiograms so the operator is able to scroll through the OCT angiogram like a cube scan. As a result, the precise location of pathology can be viewed on the corresponding OCT b-scans. This makes OCTA a better tool when detecting the exact location of a retinal pathology.

In diabetic retinopathy OCTA can show choriocapillaris abnormalities and/or retinal microvascular abnormalities such as microaneurysms, vascular remodeling adjacent to the foveal avascular zone (FAZ), enlarged FAZ, and capillary tortuosity and dilation through different stages. OCTA can show smaller vascular changes not detectable by FA.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients suffering from different stages of diabetic retinopathy.

Exclusion Criteria:

* Other ocular problems affecting vision including glaucoma, cataract, amblyopia, hypertensive retinopathy, vein occlusion and uveitis.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Mean area of FAZ in various stages of diabetic retinopathy and difference between these groups in superficial and deep capillary plexuses | baseline
  analysis of foveal avascular zone in different stages of diabetic retinopathy using OCT angiography

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Hn El Daly, MD, Study Chair — Assuit Universoty

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim DY, Fingler J, Zawadzki RJ, Park SS, Morse LS, Schwartz DM, Fraser SE, Werner JS. Optical imaging of the chorioretinal vasculature in the living human eye. Proc Natl Acad Sci U S A. 2013 Aug 27;110(35):14354-9. doi: 10.1073/pnas.1307315110. Epub 2013 Aug 5. PMID 23918361
- [Result] Choi W, Mohler KJ, Potsaid B, Lu CD, Liu JJ, Jayaraman V, Cable AE, Duker JS, Huber R, Fujimoto JG. Choriocapillaris and choroidal microvasculature imaging with ultrahigh speed OCT angiography. PLoS One. 2013 Dec 11;8(12):e81499. doi: 10.1371/journal.pone.0081499. eCollection 2013. PMID 24349078
- [Result] NOVOTNY HR, ALVIS DL. A method of photographing fluorescence in circulating blood in the human retina. Circulation. 1961 Jul;24:82-6. doi: 10.1161/01.cir.24.1.82. No abstract available. PMID 13729802